CLINICAL TRIAL: NCT04798664
Title: Comparing Smoking Cessation Interventions Among Underserved Patients Referred for Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPCC 12519
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
Keywords: Patients, Underserved; Early Detection of Cancer; Lung Cancer; Nicotine Replacement Products; Incentives; Behavioral Economics; Smoking Cessation; Nicotine Dependence
MeSH Terms: conditions — Smoking Cessation; Lung Neoplasms; Tobacco Use Disorder | interventions — Fertility

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled trial using opt-out consent with longitudinal follow-up of patients over 12 months. Based on the expected accrual at each of the four health systems, we expect that overall there will be 470 participants in basic usual care (Arm 1), and 910 participants in each of intervention arms 2-4.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Basic Usual Care (No Intervention): Participants receive the usual care approach, Ask-Advise-Refer (AAR), which is a standard approach in which non-study clinicians ask smokers about their desire to quit smoking, advise them to quit, and provide informational resources such as hotlines, specialized clinics, or smoking cessation classes.
- Enhanced Usual Care (Active Comparator): Participants receive the basic usual care of Ask-Advise-Refer as well as free access to nicotine replacement therapy (NRT) and/or reimbursement of up to $300 for any smoking cessation medications (varenicline/Chantix or bupropion/Zyban) prescribed by non-study clinicians.
  Interventions: Behavioral: Removal of Financial Barriers
- Enhanced Usual Care plus Financial Incentives (Active Comparator): Participants receive all aspects of enhanced usual care plus an incentive plan in which they will be informed of their eligibility to earn $100, $200, and $300 if they submit negative tests for nicotine metabolites at 2 weeks, 3 month and 6 months following their quit date, respectively.
  Interventions: Behavioral: Removal of Financial Barriers; Behavioral: Financial Incentives
- Enhanced Usual Care plus Financial Incentives plus Mobile Health Application (Active Comparator): Participants receive all aspects of Arm 3 plus an intervention to promote episodic future thinking (EFT), called FutureMe. EFT has been shown to reliably reduce discounting of the future. Patients will practice using EFT cues to envision the "future is now" between the time of enrollment and the quit date, and will then receive cues from the quit date through the end of the intervention period, 6 months later, unless they ask to stop receiving cues sooner.
  Interventions: Behavioral: Removal of Financial Barriers; Behavioral: Financial Incentives; Behavioral: Mobile Health Application

INTERVENTIONS:
Behavioral: Removal of Financial Barriers — Free access to nicotine replacement therapies and/or reimbursement for smoking cessation prescription medications
  Other Names: NRT
  Arms: Enhanced Usual Care; Enhanced Usual Care plus Financial Incentives; Enhanced Usual Care plus Financial Incentives plus Mobile Health Application
Behavioral: Financial Incentives — Financial incentive plan of up to $600 for biochemically-confirmed, sustained abstinence for 6 months.
  Other Names: Incentives
  Arms: Enhanced Usual Care plus Financial Incentives; Enhanced Usual Care plus Financial Incentives plus Mobile Health Application
Behavioral: Mobile Health Application — Episodic future thinking tool to overcome temporal discounting of future
  Other Names: FutureMe
  Arms: Enhanced Usual Care plus Financial Incentives plus Mobile Health Application

SUMMARY:
To compare the effectiveness of four interventions to promote sustained, biochemically confirmed smoking abstinence for 6 months among underserved smokers referred for lung cancer screening at four large U.S. health systems.

DETAILED DESCRIPTION:
We will conduct a 4-arm randomized trial comparing 4 interventions to promote sustained, biochemically confirmed smoking abstinence for 6 months among smokers in underserved demographic groups. The 3,200 participants to be enrolled will be current smokers who are Black, Hispanic, and/or have low socioeconomic status (defined as household income <200% of the federal poverty line or a high school education or less) or rural residence who are referred for low-dose computed tomography (LDCT) screening at 4 large health systems. All adult patients with LDCT orders will be further screened for eligibility. Eligible patients will enroll with opt-out consent and complete the study using the NIH-funded Way to Health online research portal. The primary outcome will be biochemically confirmed, sustained abstinence from smoking tobacco for 6 months following participants' selected quit dates. Relapse rates will be tracked at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker (≥ 1 cigarettes per day, not including e-cigarettes)
* Has a low-dose computed tomography (LDCT) scan ordered by their physician
* Underserved, defined as one or more of the following: (a) Black, (b) Hispanic, (c) rural residence, or (d) low socioeconomic status (Defined as one or both of: high-school education or less, or household income <200% of the federal poverty line)
* Able to receive study invitation and screening, by virtue of showing up to a radiology location affiliated with a participating health system for the LDCT, or having a valid email address or telephone number on file with the health system
* Access to a cell phone with text messaging or the internet
* Aged 18 years or older

Exclusion Criteria:

* No cell phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3228 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Biochemically confirmed smoking abstinence sustained for 6 months | 6 months
  The primary outcome measure is sustained abstinence for 6 months, and will require self-report of smoking cessation followed by biochemical confirmation at 2 weeks, 3, and 6 months.

SECONDARY OUTCOMES:
Quit status (self-report) | 2 weeks, 3 months, 6 months, 12 months
  Point-prevalent rates of self-reported nicotine use and tobacco product use
Quit status (biochemically confirmed) | 2 weeks, 3 months, 6 months,12 months
  Point-prevalent rates of biochemically confirmed smoking cessation
Health-related quality of life | Baseline, 6 months, 12 months
  The EuroQuol Group's quality of life (EQ-5D) scale is a 25-item validated scale used to assess patients' perceived health-related quality of life across the domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Perceived barriers to cessation | Baseline, 6 months, 12 months
  The Challenges to Stopping Smoking Scale (CSS-21) is a validated 21-item measure to assess patients' perceived barriers to smoking cessation. The CSS-21 has two sub-scales: intrinsic factors (physical, psychological or cognitive aspects of quitting) and extrinsic factors (social or environmental aspects of quitting).
Self-efficacy related to cessation efforts | Baseline, 6 months, 12 months
  We will use the 10-item situational measure of self-efficacy related to smoking behavior. This scale measures how sure participants are that they can avoid smoking in different situations.
Motivation to quit | Baseline, 6 months, 12 months
  The Stages of Change (SOC) is a validated 1-item measure to assess patient's self-reported motivation to quit.
Temporal ("delay") discounting | Baseline, 6 months, 12 months
  Temporal discounting is a measure of impulsivity that reflects people's tendencies to discount the value of a reward as a function of how far in the future it would be received. We will use the 5-Trial Adjusting Delay Task to assess temporal discounting.

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Halpern, MD PhD, Principal Investigator — University of Pennsylvania
Locations (5):
- United States (5):
  - Kaiser Permanente Southern California, Oakland, California
  - Henry Ford Health System, Detroit, Michigan
  - Geisinger, Danville, Pennsylvania
  - Lancaster General Health, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie published results will be made available to other researchers, after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months after publication and up to 36 months following publication. After 36 months the data will be available in our University's data warehouse but without support, except for deposited metadata.
Access Criteria: Proposals for data use will be reviewed by Principal Investigator and independent review board (such as the Data and Safety Monitoring Board). Approved requestors will need to sign data use agreements to access and use data.
URL: https://www.pair.upenn.edu

REFERENCES:
- [Derived] Kohn R, Vachani A, Small D, Stephens-Shields AJ, Sheu D, Madden VL, Bayes BA, Chowdhury M, Friday S, Kim J, Gould MK, Ismail MH, Creekmur B, Facktor MA, Collins C, Blessing KK, Neslund-Dudas CM, Simoff MJ, Alleman ER, Epstein LH, Horst MA, Scott ME, Volpp KG, Halpern SD, Hart JL; Stakeholder Advisory Committee. Comparing Smoking Cessation Interventions among Underserved Patients Referred for Lung Cancer Screening: A Pragmatic Trial Protocol. Ann Am Thorac Soc. 2022 Feb;19(2):303-314. doi: 10.1513/AnnalsATS.202104-499SD. PMID 34384042